CLINICAL TRIAL: NCT06692582
Title: Influence of Adjunctive Electrolysed Saline Rinse in Stage III Periodontitis Patients
Brief Title: Electrolysed Saline Rinse As an Adjunct for Treatment of Chronic Periodontitis
Acronym: EOSPERIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKCLJEOSPERIO1
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be performed using a computer program. Only one member of the research group, who will also prepare the mouthwashes, will know the content of the randomization table or the type of mouthwash used by each individual. Identification codes will remain hidden from all other researchers and subjects until the final follow-up examinations. The packaging of the mouthwashes will be identical, and the active ingredients will not be distinguishable by color.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EOS (Experimental)
  Interventions: Other: Electrolysed saline rinse
- CHX (Active Comparator)
  Interventions: Other: Electrolysed saline rinse
- Placebo - distilled water (Placebo Comparator)
  Interventions: Other: Electrolysed saline rinse

INTERVENTIONS:
Other: Electrolysed saline rinse — EOS ph = 7, 200 ppm free available Chlorine

SUMMARY:
The study will be conducted as a prospective, double-blind, parallel, randomized, placebo-controlled study at the Dental Clinic of University Medical Centre Ljubljana. It will involve a one-month test period, during which the test subjects will use either placebo, Electrolysed Oxidising Saline (EOS) or chlorhexidine (CHX) in the form of a mouthwash as an adjunct to the non-surgical treatment of chronic periodontitis (i.e. root planing and scaling). We will include 60 subjects who will be selected from consecutively scheduled patients referred by their personal dentists for periodontal treatment at the Dental Clinic of University Medical Centre Ljubljana.

DETAILED DESCRIPTION:
Before enrolment in the study, we will perform a thorough clinical examination of each patient, which will involve assessing several periodontal parameters at six sites around each tooth on all teeth, excluding third molars: plaque index (PlI), probing depth (PD), gingival recession (GR), clinical attachment loss (CAL), bleeding on probing (BOP), furcation involvement, and tooth mobility. All clinical parameters will be measured using a William's periodontal probe (Hu-Friedy, USA, PQW6). Local X-rays of sites affected by periodontitis will be taken. The performed clinical examination will not differ in any way from the examination conducted on all patients, even those not included in our study. The population of included subjects will consist of individuals of both sexes, aged 25-70 years, smokers and non-smokers, with moderate or advanced stage of chronic periodontitis (stage III, IV). They will be selected based on the following inclusion criteria: clinical attachment loss ≥ 5 mm on at least two teeth in two different jaw quadrants; presence of stable occlusion and at least 16 teeth, among which at least 12 teeth are suitable for evaluation (excluding wisdom teeth, teeth with orthodontic wires, bridges, crowns, and implants). We will exclude individuals who: suffer from chronic systemic diseases (diabetes, cancer, HIV infection, metabolic bone diseases, and diseases that interfere with wound healing processes); are undergoing radiation or chemotherapy; are taking immunosuppressants, antiepileptic drugs, calcium antagonists, nonsteroidal anti-inflammatory drugs; have been treated with antibiotics in the past 12 months; have a known allergy to CHX; have undergone scaling and root planing or surgical periodontal treatment in the past year; are pregnant or breastfeeding. Patients will be informed about the purpose of the research in writing. Prior to the commencement of the study, all patients will fill out an informed consent form.

Subjects will then be divided into three groups of 20; the first group will use a mouthwash consisting of EOS (active ingredient) for one month after the non-surgical treatment; the second group will use a mouthwash containing CHX (positive control); and the third group will use distilled water (negative control/placebo). Randomization will be performed using a computer program. Only one member of the research group, who will also prepare the mouthwashes, will know the content of the randomization table or the type of mouthwash used by each individual. Identification codes will remain hidden from all other researchers and subjects until the final follow-up examinations. The packaging of the mouthwashes will be identical, and the active ingredients will not be distinguishable by color.

Samples of subgingival fluid will be collected at the beginning of the test period for the purpose of microbiological characterization using sterile paper points from the buccal surface of four teeth (sites with the greatest probing depths in each quadrant) and transported to the laboratory of the Institute of Microbiology and Immunology using a transport medium (RTF). The microbiological analysis will be performed using Quantitative Polymerase Chain Reaction (qPCR).

Subsequently, all patients will undergo a non-surgical periodontal treatment, which will include instruction and motivation for proper oral hygiene, removal of hard and soft plaque deposits using a piezoelectric device and ultrasonic tip, and root planing and scaling under local anesthesia. Each subject will then receive a package with an identification number and the label A, B, or C on it, according to the computer-generated randomization scheme. One-third of the patients will receive EOS in the package, one-third will receive CHX, and one-third will receive distilled water. Subjects will then rinse their oral cavities with 15 ml of their allocated mouthwash twice daily (in the morning and evening) for 30 seconds for four consecutive weeks.

After four weeks, subjects will be invited for their first follow-up examination. They will report any side effects and return the packaging of the for compliance control. They will also be asked about the organoleptic properties of the mouthwash they used. We will perform a thorough clinical examination again and collect samples of subgingival fluid in the same manner as during the initial examination. The second follow-up examination will be conducted three months after the oral hygiene phase and will include a clinical assessment and collection of subgingival fluid samples.

The primary outcome variable will be the number of residual diseased sites (PD > 4mm + BOP). Secondary outcome variables will include plaque index assessment, BOP, PD, and quantity of periodontopathogens. Since teeth are "nested" within patients and probing sites are "nested" within teeth, the collected data is interdependent. A multilevel multiple logistic regression model will therefore be used to examine associations between variables.

ELIGIBILITY:
Inclusion Criteria:

Clinical attachment loss ≥ 5 mm on at least two teeth in two different jaw quadrants; presence of stable occlusion and at least 16 teeth, among which at least 12 teeth are suitable for evaluation (excluding wisdom teeth, teeth with orthodontic wires, bridges, crowns, and implants).

Exclusion Criteria:

We will exclude individuals who: suffer from chronic systemic diseases (diabetes, cancer, HIV infection, metabolic bone diseases, and diseases that interfere with wound healing processes); are undergoing radiation or chemotherapy; are taking immunosuppressants, antiepileptic drugs, calcium antagonists, nonsteroidal anti-inflammatory drugs; have been treated with antibiotics in the past 12 months; have a known allergy to CHX; have undergone scaling and root planing or surgical periodontal treatment in the past year; are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
No of residual diseased sites | Baseline, 1 month, 3 months
  Probing Pocket Depth (PPD) > 4 mm + Bleeding On Probing (BOP)

SECONDARY OUTCOMES:
Probing Pocket Depth (PPD) | Baseline, 1 month, 3 months
Clinical Attachment Level (CAL) | Baseline, 1 month, 3 months
Full Mouth Plaque Score (FMPS) | Baseline, 1 month, 3 months

OTHER OUTCOMES:
Absolute number and share of 14 periodontopathogenic species | Baseline, 1 month, 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided